CLINICAL TRIAL: NCT03332693
Title: Macroscopic and Molecular Changes in Knee Muscular - Tendon Unit in Response to Acute Resistant Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HYMC-0058-16
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Physical Exertion
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No exercise (Active Comparator): Volunteers will not participate in exercise
  Interventions: Other: No exercise
- Light exercise (Active Comparator): Volunteers will participate in one short exercise
  Interventions: Other: Exercise
- Heavy exercise (Active Comparator): Volunteers will participate in heavy exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Leg weight raising
  Arms: Heavy exercise; Light exercise
Other: No exercise — Volunteers will not participate in exercise
  Arms: No exercise

SUMMARY:
The aim of this study is to determine whether individuals differ one from the other in their genetic, cellular, systemic, structural and functional response to acute exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Unhealthy adults

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphism changes in knee muscles | One year
  Genetic analysis will be made through a blood test and biopsy of knee muscle and results will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Eias Kassem, MD, Study Director — Hillel Yaffe Medical Center; Sigal Ben Zaken, PhD, Principal Investigator — Wingate Academic College for Physical Education and Sport Sciences
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel